CLINICAL TRIAL: NCT04474379
Title: Prospective Memory Impairment in Parkinson Disease-related Cognitive Decline: Intervention and Mechanisms
Brief Title: Everyday Memory Impairment in PD-related Cognitive Decline
Acronym: PMT2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Erin Foster, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202007054
Record Dates: First submitted 2020-07-10; First posted 2020-07-16 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction | interventions — Time

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to treatment arm (1:1 ratio, stratified by sex and Clinical Dementia Rating (CDR) Score 0 or 0.5): the strategy training or the process training.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and outcomes assessor will be blind to which cognitive training a participant will be randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strategy Training (Experimental): Consists of 8-90 minute sessions over 8 weeks. In sessions 1 and 2, in addition to teaching about event- and time-based tasks, the therapist teaches the participant specific strategies for each type of task (implementation intentions for event-based and strategic clock-checking for time-based) and instructs in their use before and during the training games. In sessions 3-8, the tester tells the participant s/he will be practicing both types of tasks in the training games and can support the participant's strategy use if needed. Feedback on accuracy and strategy use are provided after each training game. After completing the training games, the therapist and participant discuss how the strategies can be applied to the participant's real-life prospective memory goals, and the therapist helps the participant develop written action plans to do so. Plans and goals are reviewed and modified, if necessary, at each session.
  Interventions: Behavioral: Strategy Training (Time- and Event- Based)
- Process Training (No Intervention): Consists of 8, 90 minute sessions over 8 weeks. In sessions 1 and 2, the therapist teaches the participant about event- and time-based prospective memory tasks, respectively. In sessions 3-8, the tester tells the participant that s/he will be practicing both types of tasks in the training games. In all sessions, the participant completes the training games with no strategy instruction from the therapist. Feedback on accuracy is provided after each training game. This is typical of a process training approach and expects that practice of the training tasks will improve prospective memory ability per se or that participants will develop effective strategies for completing prospective memory tasks on their own. At the end of each session, the therapist reminds the participant of his/her real-life prospective memory goals, provides a handout that lists the goals, and instructs the participant to try to complete them as intended. Goals are reviewed and modified if necessary.

INTERVENTIONS:
Behavioral: Strategy Training (Time- and Event- Based) — In time-based training, strategic clock-checking behavior is taught by requiring participants to click a button to reveal the virtual time of day. Event-based training involves implementation intention methods.
  Arms: Strategy Training

SUMMARY:
The investigators will aim enroll participants into our study within 3-6 months after their parent study visit so the investigators can utilize some key data points (e.g. PD-MCI diagnosis, rs-fcMRI data) from that study. PD participants will participate in a single-blind RCT with two treatment arms: process training and strategy training (Fig 4). They will complete pre-training assessment (Pre), be randomized to treatment arm (1:1 ratio stratified by sex), and then complete 8 training sessions over an 8-week period. They will return within 1 week for post-training assessment (Post) and then will complete Follow-up (FU) assessments via web or mailed survey 3 and 6 months after training ends. They will complete a 12mo FU assessment in person in conjunction with their annual parent study visit. HC participants will complete prospective memory assessment at one time point coinciding with (or within 3-6 months of) their parent study visit to determine whether any relationships observed between rs-fcMRI data and prospective memory are specific to PD.

DETAILED DESCRIPTION:
Parkinson disease (PD) causes cognitive deficits that can impair instrumental activities of daily living function and quality of life (QOL) even in the absence of dementia. Currently, there are no treatments to address this pressing burden and, even worse, some medical treatments for PD can exacerbate cognitive deficits. For these reasons, behavioral interventions that attenuate the negative functional consequences of cognitive decline in PD and thus potentially delay the onset of dementia are in high demand. An intervention that enables people with PD to remember to perform necessary and meaningful daily activities could improve or maintain their independence, disease self-management, participation in society, and reduce caregiver burden. The primary goal of this study is to determine the efficacy of such an intervention. Importantly, in doing so, the investigators will directly address a critical point of contention in cognitive intervention research: Which approach (process or strategy training) is the best option for producing functionally-relevant benefits for people with PD? Additionally, the study team will investigate behavioral and neurobiological correlates of prospective memory in PD, including individual characteristics that may predict treatment response. This work will lead to a targeted and tailored biobehavioral intervention that optimizes function, promotes QOL, and improves the long-term management of a common chronic neurological condition. It will move the field of rehabilitation forward by providing valuable theoretical and practical information related to the type of cognitive intervention approach that is most appropriate for people with PD. This then will stimulate and justify the channeling of future research efforts and funding toward further development, testing, dissemination, and implementation of said approach.

Primary Outcomes:

Aim 1. Laboratory prospective memory performance - The Virtual Week test will be administered to PD participants at Pre and Post to assess near transfer of training objectively (primary endpoint). It will also be administered to PD participants at 12mo FU to explore long term training effects (secondary endpoint) and to HC participants at Pre to investigate neural mechanisms of prospective memory performance (Aim 3). It is a computerized board game that simulates daily life and real-world prospective memory challenges. Each circuit represents one day in which the participant completes time-appropriate activities and makes choices about them. Embedded in each day are 8 prospective memory tasks (4 event, 4 time). Participants complete a practice day and then 4 test days; equivalent versions are counterbalanced across testing sessions. The main outcome variable is prospective memory accuracy, defined as the proportion of correct prospective memory responses (32 total: 16 event, 16 time). To further explore the effects of time-based training, the investigators will record strategic clock-checking behavior by requiring participants to click a button to reveal the virtual time of day.

Aim 2. Reported everyday prospective memory: (2a) General everyday prospective memory function - The Prospective and Retrospective Memory Questionnaire (PRMQ)will be administered via web-based or mailed survey to PD participants and informants at Pre, Post and 3mo FU to assess far transfer of training (primary endpoint), to PD participants and informants at 6mo and 12mo FU to explore long term training effects (secondary endpoint), and to HC participants at Pre to determine neural mechanisms of everyday prospective memory (Aim 3). The PRMQ is the most widely used questionnaire for everyday prospective memory. Participants rate the frequency of 8 everyday prospective memory failures (1=Never, 5=Very Often), item scores are summed, and higher scores indicate worse everyday prospective memory. The PRMQ includes environment- and self-cued subscales (4 items each) that parallel the event- and time-based task distinction, respectively. (2b) Personalized real-life prospective memory tasks - The Bangor Goal-Setting Interview (BGSI)offers a standardized means of eliciting individual goals and rating goal attainment over time and has been successfully used in cognitive rehabilitation RCTs with older adults, including those with mild to moderate dementia. During the first two training sessions, after an explanation of the prospective memory task types (session 1: event, session 2: time), participants will complete the BGSI with the trainer to identify and set goals for 3-6 real-life prospective memory tasks they anticipate having to complete over the training period. They and their informants will rate their Pre and Post attainment of these goals on a 10-point scale (1=never remember to do; 10=always remember to do). Goal attainment ratings are averaged to yield mean attainment scores.

Additional measures:

Aims 3 & 4. Neural correlates of prospective memory and treatment response - Rs-fcMRI data will be collected and managed under the auspices of the parent study at Pre. Briefly, MRIs will be completed OFF PD medications on a 3T Siemens Prisma scanner with a 20 channel head coil and include up to 6 BOLD rs-fcMRI scans (416 volumes/run, TE=26.6ms, TR=800ms, FOV= 213mm, flip angle=61°, 3mm3 voxels; multiband factor=4; 5:39min) during fixation (eyes open). More details, including rigorous quality control methods, are in references. The investigators will use a network-level analysis approach using standard nodes from canonical networks. Our primary variables of interest will be intranetwork integrity scores, calculated based on the cross-correlations of each node within the network, for the following cognitive networks: DMN, CON, FPN, PMN, and MTL. Alternate approaches may include seed-based analyses (e.g. DLPFC) and Object Oriented Data Analysis followed by post-hoc identification of significant networks.

Aim 4. Behavioral predictors of treatment response - Based on our pilot RCT (Prelim Data 2)1, The investigators will administer the Credibility and Expectancy Questionnaire (CEQ) and Beck Depression Inventory-II (BDI-II) at Pre as potential motivational predictors of treatment response. The CEQ will be administered at the end of training session 2, so participants have some knowledge of the intervention on which to base their perceptions of credibility and expectancy. The investigators will utilize the extensive neuropsychological data collected at Pre in the parent study to assess potential cognitive predictors of treatment response. Our primary cognitive variables will be the domain z-scores for Memory and Executive Function, computed as the average of standardized scores from measures assessing that domain. Other - PD (and normal cognition for HCs) will be determined via MDS Level II diagnostic criteria in the parent study based on a comprehensive neuropsychological assessment battery and in-depth clinical interviews (CDR). In addition to the main measures of interest described above, the investigators will collect other data to characterize participants, as covariates, or as secondary outcomes (Table 3). This will permit exploration of the influence of sex or other relevant biological variables (e.g. co-morbidities, medication) and broader functional outcomes. The investigators will obtain much of this data from the parent study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over age 50 who meet criteria for typical idiopathic PD
* Hoehn & Yahr stage I-III,
* Treated with levodopa/carbidopa
* Have subjective memory complaints (as identified in phone screen),
* Have an informant to complete relevant ratings,
* Medications should be stable for 4 weeks prior with no changes planned during the treatment portion of the study (Pre to Post); changes over the follow-up period will be tracked and accounted for as appropriate.

Exclusion Criteria:

* Dementia according to MDS criteria or MoCA score <21.
* Other neurological disorders (e.g. stroke, seizures), brain surgery, severe systemic diseases, major psychiatric disorder or history of psychotic symptoms (e.g. schizophrenia, bipolar disorder, delusions, hallucinations), or drug abuse.
* Treatment with medications that interfere with cognition (e.g. anticholinergics).
* Any other condition that would interfere with participation (e.g., non-English speaking, significant current depression).
* Psychiatric conditions/ symptoms that are common in PD (e.g. anxiety, depression) are allowed if they are deemed insufficient to interfere with participation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Virtual Week Computer-based Memory Test performance after 5-weeks and 12-month post-intervention. | Administered at baseline, pre-treatment session; One week post-treatment (approximately five weeks after the baseline test); and 12-months post-strategy training sessions.
  A computer-based prospective memory test that simulates a real day where a person has to remember to do tasks.
Change in The Prospective and Retrospective Memory Questionnaire scores after 5-weeks, 3-months, 6-months, and 12-month post-intervention. | Administered at baseline, pre-treatment session; One week post-treatment (approximately five weeks after the baseline test); then 3-, 6- and 12-months post-completion of strategy training sessions.
  Participant-reported everyday prospective memory
Change in Bangor Goal Setting Interview goal attainment after 5-weeks and 12-month post-intervention. | Administered at baseline, pre-treatment session; One week post-treatment (approximately five weeks after the baseline test); and 12-months post-strategy training sessions.
  A standardized measure that elicits individual goals and rating goal attainment over time

CONTACTS AND LOCATIONS:
Overall Officials: Erin Foster, PhD, OTD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD that underlie results in a publication. Unpublished data may be shared at the PI's discretion. All shared data will be deidentified.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 3 months after publication
Access Criteria: Per individual request to PI.